CLINICAL TRIAL: NCT01206335
Title: A Phase II Open Label Study With OHR/AVR118 in Anorectic Patients With Recurrent or Advanced Malignancies
Brief Title: Open Label Study With OHR/AVR118 in Advanced Cancer Patients With Anorexia-Cachexia
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ohr Pharmaceutical Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OHR-201
Record Dates: First submitted 2010-09-20; First posted 2010-09-21 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Anorexia; Cancer Cachexia
Keywords: Cancer Cachexia; Anorexia; Advanced Malignancies; Weight Loss; Fatigue; Karnofsky; C-Reactive Protein; Simmonds Functional Assessment
MeSH Terms: conditions — Anorexia; Weight Loss; Fatigue | interventions — EOM613

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- OHR/AVR118 (Experimental): Experimental Drug
  Interventions: Drug: OHR/AVR118

INTERVENTIONS:
Drug: OHR/AVR118 — OHR/AVR118 given subcutaneously at 4mL per day
  Other Names: AVR118

SUMMARY:
The purpose of this study is to determine whether patients with advanced cancers who receive OHR/AVR118 solution for injection into the skin can achieve improvement in quality of life. Based on a previous study in patients with AIDS, possible benefits may include improved appetite and strength; weight gain, improved mood; and decreased fatigue.

DETAILED DESCRIPTION:
Advanced cancers are usually debilitating. There are few treatments available for symptoms of advanced cancers like loss of appetite, decreased strength, fatigue, and change in mood. This Phase II, open label study with OHR/AVR118 will enable the Sponsor to gather data on safety and efficacy of OHR/AVR118 in the patient population with anorexia-cachexia. Patients aged 18-85 with advanced cancers (excluding central nervous system [CNS] cancers) who may or may not be receiving chemotherapy, may be eligible to participate. The study drug, 4.0 mL, will be given subcutaneously each day for 28 days. Patients who respond to the trial period dosing will be eligible to continue on OHR/AVR118 if they and their physicians believe it would be beneficial, and if no safety concerns are raised.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor cancer, leukemia, lymphoma, or multiple myeloma.
* Concurrent anti-cancer treatment, such as chemotherapy or radiation therapy is permitted except for neo-adjuvant or adjuvant programs.
* Between the ages of 18-85.
* Symptoms of recurrent or metastatic cancer in which anorexia is a predominant symptom, not necessarily associated with cachexia, and are not attributed to anemia, concomitant illnesses, or obstruction or loss of organ function.
* Karnofsky performance status of 40%
* Palliative Prognostic Score (PaP) of less than 6
* Patient is expected to be able to remain on a study protocol for two months.
* Pretreatment laboratory data within 7 days of enrollment:
* Hemoglobin >8.5 g/dL , or on stable doses (hematocrit stable within 1 gram and dose stable for one month) of erythropoietin or similar medication.
* Absolute neutrophil count (ANC) 1,500/mm3.
* Platelets 50,000/mm3.
* Total bilirubin 2.0
* ALT and AST 2.5 times the ULN, or, if the patient has liver metastases, 5 times the ULN.
* Creatinine 1.5 mg/dL.
* Normal TSH
* Testosterone levels determined.
* Voluntary written informed consent before performance of any study-related procedure that is not part of normal medical care.
* Ability to self-administer subcutaneous medication if an assistant or nurse is not available, and to keep a compliance journal documenting injections at home.
* If on an antidepressant, the dose must have been stabilized for at least 30 days.
* Female patient is post-menopausal, surgically sterilized, or willing to use acceptable methods of birth control (i.e., a hormonal contraceptive, intra-uterine device, diaphragm with spermicide, or condom with spermicide, or abstinence) for the duration of the study.
* Male patient agrees to use an acceptable barrier method for contraception during the study

Exclusion Criteria:

* Patient has uncontrolled brain metastases or central nervous system disease.
* Patient has mechanical, non-reversible reason for not being able to eat, or have a potential for developing malignant bowel obstruction during the course of the induction phase of treatment, or patients requiring a PEG for obstruction.
* Patient has had any major surgery within four weeks of enrollment.
* Patient has an uncontrolled concomitant illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, or cardiac arrhythmia.
* In the Investigator's opinion, potentially interfere with the completion of treatment according to this protocol.
* Female patient is pregnant or breast-feeding.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2010-09; Primary Completion 2012-12 (Estimated); Study Completion 2013-02 (Estimated)

PRIMARY OUTCOMES:
Alleviation of multiple cachexia symptoms | Four weeks
  Functional Status/Quality of Life as assessed by Simmonds Functional Assessment (SFA); Appetite and early satiety as assesed by patetient-generated subjective global assessment (PG-SGA), Edmonton Symptom assessment Scale (ESAS) and dyspepsia symptom severity index (DSSI); weight gain; increase in lean body mass.

SECONDARY OUTCOMES:
Impact on inflammatory markers and hormonal milieu | 4 weeks
  Measurement of effects on Testosterone, TSH and C-Reactive protein

CONTACTS AND LOCATIONS:
Overall Officials: Martin Chasen, MBChB, Principal Investigator — Ottawa Hospital Cancer Centre
Locations (1):
- Ottawa Hospital Cancer Centre, Ottawa, Ontario, Canada